CLINICAL TRIAL: NCT03305562
Title: Pediatric Hypertension Registry (PHREG)
Acronym: PHREG
Status: Terminated | Type: Observational
Why Stopped: Study was a pilot study and the investigators received funding to initiate the main study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00046001
Record Dates: First submitted 2017-09-27; First posted 2017-10-10 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Hypertension; Pediatric Disorder
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The cohort of patients seen prior to the implementation of a standardized clinical management protocol on 10/01/2017 whose data is collected retrospectively.
- Prospective cohort: The cohort of patients seen initially seen after implementation of a standardized clinical management protocol on 10/01/2017 whose data is collected prospectively.

SUMMARY:
Pediatric hypertension is increasingly common and is a precursor for adult cardiovascular and renal disease. But even during childhood, hypertension is associated with significant morbidity, including cognitive impairment and organ damage. However, the cause of pediatric hypertension, the response to treatment, and the mechanisms behind organ damage are incompletely understood. Due to these limitations, there are no first-line medications, and treatment is often inadequate. An improved comprehension of the course of pediatric hypertension could enhance clinical care. The goal of this proposal is to create a registry of patients with hypertension to better enable research into this important disease. This patient registry will enhance the investigators ability to quickly collect and analyze data for research studies.

DETAILED DESCRIPTION:
The investigators will include all subjects evaluated at the Brenner Children's Hospital Pediatric Nephrology clinic since January 1st, 2013 with a diagnosis of high blood pressure confirmed with three separate blood pressure measurements >=90th percentile for age, sex, and height, or >120/80 mmHg. The investigators will exclude patients whose initial evaluation occurred on or after their 18th birthday.

ELIGIBILITY:
Inclusion Criteria:

- Patients at one of the following : Wake Forest Baptist Health Brenner Children's Hospital Pediatric Nephrology clinic Emory University Pediatric Nephrology

* Diagnosis of hypertension confirmed with three separate blood pressure measurements
* Diagnosis after January 2013
* >90th percentile for age, sex, height, or >120/80.

Exclusion Criteria:

- Patients whose initial evaluation occurred on or after their 18th birthday.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects that are patients in the Brenner Children's Hospital Pediatric Nephrology Clinic or Emory University Pediatric Nephrology with a confirmed diagnosis of high blood pressure.
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 10 years
  Auscultated blood pressure measurements in clinic
Left ventricular hypertrophy | 10 years
  Left ventricular hypertrophy and other cardiac structural/function changes on echocardiograms
Albuminuria | 10 years
  Urinary albumin-to-creatinine (>30 mg/g)

SECONDARY OUTCOMES:
Ambulatory blood pressure | 10 years
  Ambulatory blood pressure monitoring data
Renal function | 10 years
  Glomerular filtration rate
Uric acid | 10 years
  Serum uric acid

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M South, MD MS, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Emory University Pediatric Nephrology, Atlanta, Georgia
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Din-Dzietham R, Liu Y, Bielo MV, Shamsa F. High blood pressure trends in children and adolescents in national surveys, 1963 to 2002. Circulation. 2007 Sep 25;116(13):1488-96. doi: 10.1161/CIRCULATIONAHA.106.683243. Epub 2007 Sep 10. PMID 17846287
- [Background] Richey PA, Disessa TG, Somes GW, Alpert BS, Jones DP. Left ventricular geometry in children and adolescents with primary hypertension. Am J Hypertens. 2010 Jan;23(1):24-9. doi: 10.1038/ajh.2009.164. Epub 2009 Oct 22. PMID 19851297
- [Background] King JT Jr, DiLuna ML, Cicchetti DV, Tsevat J, Roberts MS. Cognitive functioning in patients with cerebral aneurysms measured with the mini mental state examination and the telephone interview for cognitive status. Neurosurgery. 2006 Oct;59(4):803-10; discussion 810-1. doi: 10.1227/01.NEU.0000232666.67779.41. PMID 17038944
- [Background] Washburn LK, Nixon PA, Russell GB, Snively BM, O'Shea TM. Preterm Birth Is Associated with Higher Uric Acid Levels in Adolescents. J Pediatr. 2015 Jul;167(1):76-80. doi: 10.1016/j.jpeds.2015.03.043. Epub 2015 Apr 11. PMID 25868431
- [Background] Feig DI, Soletsky B, Johnson RJ. Effect of allopurinol on blood pressure of adolescents with newly diagnosed essential hypertension: a randomized trial. JAMA. 2008 Aug 27;300(8):924-32. doi: 10.1001/jama.300.8.924. PMID 18728266
- [Background] Mazzali M, Hughes J, Kim YG, Jefferson JA, Kang DH, Gordon KL, Lan HY, Kivlighn S, Johnson RJ. Elevated uric acid increases blood pressure in the rat by a novel crystal-independent mechanism. Hypertension. 2001 Nov;38(5):1101-6. doi: 10.1161/hy1101.092839. PMID 11711505
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Schwartz GJ, Brion LP, Spitzer A. The use of plasma creatinine concentration for estimating glomerular filtration rate in infants, children, and adolescents. Pediatr Clin North Am. 1987 Jun;34(3):571-90. doi: 10.1016/s0031-3955(16)36251-4. PMID 3588043
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Khoury PR, Mitsnefes M, Daniels SR, Kimball TR. Age-specific reference intervals for indexed left ventricular mass in children. J Am Soc Echocardiogr. 2009 Jun;22(6):709-14. doi: 10.1016/j.echo.2009.03.003. Epub 2009 May 7. PMID 19423289
- [Background] Rademacher ER, Sinaiko AR. Albuminuria in children. Curr Opin Nephrol Hypertens. 2009 May;18(3):246-51. doi: 10.1097/MNH.0b013e3283294b98. PMID 19276802

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03305562/Prot_002.pdf
  • Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03305562/ICF_001.pdf